CLINICAL TRIAL: NCT01926548
Title: Open-label, Randomized, Single-dose, 2-way Crossover Study to Evaluate the Pharmacokinetics(Cmax, Auc) of CJ Imatinib Mesylate Tablet 200mg x 1 Compared With Gleevec Film-coated Tablet 100mg x 2 in Healthy Male Volunteers
Brief Title: to Evaluate the Pharmacokinetics(Cmax, Auc) of CJ Imatinib Mesylate Tablet 200mg x 1 Compared With Gleevec Film-coated Tablet 100mg x 2 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_IMM_101
Record Dates: First submitted 2013-08-14; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety

ARMS (2):
- CJ Imatinib 200mg (Experimental): 1 tablet(200mg) a day,PO,QD
  Interventions: Drug: CJ Imatinib mesylate tablet
- Gleevec 100mg (Active Comparator): 2 tablet(100mg) a day,PO,QD
  Interventions: Drug: Gleevec film-coated tablet 2 x 100mg

INTERVENTIONS:
Drug: CJ Imatinib mesylate tablet
  Arms: CJ Imatinib 200mg
Drug: Gleevec film-coated tablet 2 x 100mg
  Arms: Gleevec 100mg

SUMMARY:
This study is designed to evaluate the pharmacokinetics of CJ Imatinib mesylate tablet 1 x 200mg compared with Gleevec film-coated tablet 2 x 100mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 55 years old
* Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data
* Body Mass Index (BMI) in the range of 18.5 to 27 kg/m2
* Available for the entire study period
* Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

* History of clinically significant hepatic, renal, neurology, psychiatric, pulmonary, endocrine, hematologic, cardiovascular disease
* Clinically significant vital sign

  * SBP(Systolic Blood Pressure) ≤ 90 mmHg or SBP ≥ 140 mmHg
  * DBP(Diastolic Blood Pressure) ≤ 60 mmHg or DBP ≥ 100 mmHg
* History of surgery except or gastrointestinal disease which might significantly change absorption of medicines
* History of clinically significant allergies, including imatinib
* Clinical laboratory test values are outside the accepted normal range

  * AST(ASpartate Transaminase), ALT(ALanine Transaminase)( > 1.5 times to normal range
  * Estimated GFR(Glomerular Filtration Rate) < 80 mL/min
* History of caffeine, alcohol, smoking abuse

  * caffeine > 4 cups/day
  * grapefruit juice > 4 cups/day
  * smoking > 20 cigarettes/day
  * alcohol > 140g/week
* Participated in a previous clinical trial within 3 months prior to dosing
* Donated blood within 60 days prior to dosing
* Use of prescription only medicine and oriental medicine within the 14 days before dosing or use of non-prescription medicine within the 10 days before dosing
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
maximum concentration, Area under the concentration-time curve from zero to infinity | Blood sampling up to 72hs post dose(16 times).
  Administration of IP : 1day

SECONDARY OUTCOMES:
Time to peak concentration, t1/2, Area under the concentration-time curve from zero to infinity | Blood sampling up to 72hs post dose(16 times).
  Administration of IP : 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea